CLINICAL TRIAL: NCT00080483
Title: Will Testosterone and Growth Hormone Improve Bone Structure?
Brief Title: Testosterone and Growth Hormone for Bone Loss in Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Peter Snyder, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR050618 (NIH); R01AR050618 (NIH); NIAMS-118
Record Dates: First submitted 2004-04-05; First posted 2004-04-06 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2013-12

CONDITIONS: Hypopituitarism; Hypogonadism; Growth Hormone Deficiency
MeSH Terms: conditions — Hypopituitarism; Hypogonadism; Dwarfism, Pituitary | interventions — Testosterone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Testosterone transdermally 5 g a day and somatropin subcutaneously 2 µg/kg body weight a day
  Interventions: Drug: Testosterone plus somatropin
- 2 (Active Comparator): AndroGel transdermally 5 g a day for two years
  Interventions: Drug: testosterone

INTERVENTIONS:
Drug: Testosterone plus somatropin — AndoGel 5 grams transdermally a day for two years Somatropin 2 µg/kg body weight/day for two years
  Arms: 1
Drug: testosterone — AndroGel transdermally 5 g a day for two years
  Arms: 2

SUMMARY:
Deficiency of testosterone, growth hormone, or both hormones can result in osteoporosis. If either hormone is replaced, the condition of the bones improves. The purpose of this study is to determine if dual hormone treatment for men deficient in testosterone and growth hormone improves bone structure more than testosterone treatment alone.

DETAILED DESCRIPTION:
Replacement of testosterone or growth hormone in patients who are deficient improves osteoporosis associated with these deficiencies. In some tissues, such as muscle, the effects of testosterone and growth hormone are additive, but it is not known if the effects are additive in bone as well. This study will compare the effects of testosterone alone with testosterone plus growth hormone in improving bone structure in men with total pituitary hormone deficiency.

Participants in this study will be men who have pituitary or hypothalamic disease and have deficiencies of all pituitary hormones, but who have not been treated with either testosterone or growth hormone. The men will be randomly assigned to receive either testosterone alone or testosterone plus growth hormone for two years. Testosterone in a gel form will be applied daily to the skin. Growth hormone will be self-administered by daily subcutaneous injection. Blood concentrations of both hormones will be monitored with blood tests every 3 months during the 2-year study. Doses of the hormones will be adjusted to keep blood concentrations of the hormones within the normal range. Changes in bone structure will be assessed noninvasively before treatment and after one year and two years of treatment by magnetic resonance microimaging (µMRI) and dual energy X-ray absorptiometry (DEXA).

ELIGIBILITY:
Inclusion Criteria:

* Documented hypothalamic or pituitary hormone deficiency
* Testosterone deficiency, defined as total serum testosterone less than 250 ng/dL at two 8 AM readings
* Growth hormone deficiency, defined by either of the following:
* For subjects who have thyroxine and cortisol deficiencies, either a subnormal age-specific IGF-1 or a peak GH response to arginine-GHRH of less than 4.1 ng/mL
* For subjects who do not have thyroxine and cortisol deficiencies, either a subnormal age-specific IGF-1 or a peak GH response to arginine-GHRH of less than 4.1 ng/mL
* Duration of testosterone and growth hormone deficiencies of two years or more
* Replacement of cortisol and/or thyroxine deficiencies
* Able to give informed consent

Exclusion Criteria:

* Current testosterone treatment or treatment during the two years prior to study entry
* Current growth hormone treatment or treatment during the three years prior to study entry
* Use of other prescription or over-the-counter androgens (androstenedione, DHEA), estrogens, or antiandrogens (spironolactone, ketoconazole)
* Diseases that could influence bone, such as hyperparathyroidism
* Medications that could influence bone, such as anticonvulsants or glucocorticoids (prednisone greater than 20 mg/day for longer than 2 weeks/year). Calcium and over-the-counter vitamin D supplements are allowed.
* Cancer that could limit life expectancy to fewer than 5 years
* Neuromuscular disease or history of stroke with residual neurological defect
* Severe or uncontrolled psychiatric illness or dementia
* Noncancerous enlargement of the prostate gland (American Urological Association symptom score greater than 21)
* Prostate cancer by history, prostate nodule on digital rectal exam (DRE), or prostate specific antigen (PSA) greater than 4
* Current alcohol or drug dependence
* Heart failure (New York class III or IV)
* Unstable angina
* Myocardial infarction within 3 months of study entry
* Liver disease (ALT greater than 3 x normal)
* Renal disease (serum creatinine greater than 2.5 mg/dl)
* Diabetes mellitus (glycosolated hemoglobin greater than 8.0%)
* Hypertension (systolic BP greater than 160 or diastolic BP greater than 100 mm Hg)
* Hematocrit greater than 48%
* Weight greater than 300 pounds
* Poor quality scan at baseline even when repeated
* Untreated, severe, obstructive sleep apnea (Epworth sleepiness score greater than 10)
* Unable to undergo an MRI because of a cardiac pacemaker or ferrometallic objects in the body

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Snyder, MD, Principal Investigator — University of Pennsylvania; Cecilia Lansang, MD, Principal Investigator — University of Florida
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Al Mukaddam M, Rajapakse CS, Bhagat YA, Wehrli FW, Guo W, Peachey H, LeBeau SO, Zemel BS, Wang C, Swerdloff RS, Kapoor SC, Snyder PJ. Effects of testosterone and growth hormone on the structural and mechanical properties of bone by micro-MRI in the distal tibia of men with hypopituitarism. J Clin Endocrinol Metab. 2014 Apr;99(4):1236-44. doi: 10.1210/jc.2013-3665. Epub 2014 Jan 13. PMID 24423356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was initiated in December, 2004 and enrollment ended in September 2008. Forty nine subjects were screened; 14 were screen failures and 35 subjects were randomized. Four subjects were withdrawn and 31 subjects completed the study.
Groups:
- 1Testosterone Only: Testosterone transdermally 5 g a day
- 2Testosterone Plus Growth Hormone: AndroGel transdermally 5 g a day somatropin subcutaneously 2 µg/kg body weight a day
Period: Overall Study
Arm/Group | 1Testosterone Only | 2Testosterone Plus Growth Hormone
Started | 17 | 18
Completed | 15 | 16
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1Testosterone Only | 2Testosterone Plus Growth Hormone | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 18 | 35
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: MicroMRI-derived Structural (Bone Volume Fraction-BVF) of the Distal Tibia at Baseline and After One and Two Years of Treatment.
Description: Increased bone volume fraction (the fraction of bone that is bone, as opposed to the fraction that is marrow), as determined by magnetic resonance of the distal tibia
Time Frame: baseline, one year, two years
Population: All subjects who had both baseline and one year evaluations
Measure: Mean (Standard Error); unit: unitless
Groups:
- 1 The Effects of Testosterone Combined With G: AndroGel transdermally 5 g a day and somatropin subcutaneously 2 µg/kg body weight a day
  AndroGel plus somatropin: AndoGel 5 grams transdermally a day for two years Somatropin 2 µg/kg body weight/day for two years
- 2 The Effects of Testosterone Alone on Structural and Mechanic: AndroGel transdermally 5 g a day for two years
  testosterone: AndroGel transdermally 5 g a day for two years
Arm/Group | 1 The Effects of Testosterone Combined With G | 2 The Effects of Testosterone Alone on Structural and Mechanic
Number analyzed (Participants) | 17 | 15
unitless
  baseline | 0.112 (0.004) | 0.104 (0.004)
  one year | 0.119 (0.004) | 0.111 (0.006)
  two years | 0.123 (0.005) | 0.114 (0.005)

2. Other Pre Specified Outcome: Increased Trabecular Thickness, as Determined by Magnetic Resonance of the Distal Tibia
Time Frame: 2 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Improved Architectural Parameters of Trabecular Bone Reflecting Connectivity, as Determined by Magnetic Resonance Imaging
Time Frame: 2 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Increased Cortical Thickness and Cortical Density, as Determined by Peripheral Quantitative Computed Tomography of the Tibial Metaphysis
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse events were reported for the 32 subjects who completed one or more years of the study.
Arm/Group | 1Testosterone Only | 2Testosterone Plus Growth Hormone
Serious Adverse Events (participants affected / at risk) | 4/17 | 4/18
Other Adverse Events (participants affected / at risk) | 10/17 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1Testosterone Only (N=17) | 2Testosterone Plus Growth Hormone (N=18)
cholycystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
coronary artery disease (Cardiac disorders) | 1 (2) | 0 (0) — stent insertion
sellar mass (Nervous system disorders) | 1 (1) | 1 (1) — transphenoidal surgery for sight increase in sellar mass
memory loss (Nervous system disorders) | 1 (1) | 0 (0) — hospitalization for observation due to brief memory loss
arthritis of knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — knee replacement
fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cancer of prostate (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1Testosterone Only (N=17) | 2Testosterone Plus Growth Hormone (N=18)
fatigue (General disorders) | 1 (1) | 2 (2)
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
increase in blood pressure (Cardiac disorders) | 1 (1) | 1 (1)
tooth infection (Infections and infestations) | 2 (4) | 0 (0)
hypothyroid (Endocrine disorders) | 2 (2) | 3 (3)
constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (9)
anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
elevated PSA (Reproductive system and breast disorders) | 1 (1) | 3 (3)
positive Tinnel's sign (Nervous system disorders) | 0 (0) | 4 (4)
headache (Nervous system disorders) | 0 (0) | 2 (2)
urinary tract infection (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No